CLINICAL TRIAL: NCT06567119
Title: A Randomized, Double-blind, Placebo-controlled Exploratory Clinical Study to Evaluate the Safety and Tolerability of SPOT-mRNA01 Injection in Healthy Adult Subjects.
Brief Title: Preliminary Evaluation of the Safety and Tolerability of SPOT-mRNA01 Subcutaneously Administered in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SIPO Biotechnology Co. Ltd. (Industry)
Collaborators: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FM-T1-SH; NCT06438341 (obsolete NCT alias)
Record Dates: First submitted 2024-08-14; First posted 2024-08-22 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Skin Aging
Keywords: SPOT-mRNA01; COL1A1 mRNA; EVs

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPOT-mRNA01 (Active Comparator): SPOT-mRNA01 (COL1A1 mRNA-loaded by EVs)
  Interventions: Biological: SPOT-mRNA01
- Placebo (Placebo Comparator): Sterile isotonic solution
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: SPOT-mRNA01 — SPOT-mRNA01 (COL1A1 mRNA-loaded by EVs) ,single-dose subcutaneous injection
  Arms: SPOT-mRNA01
Other: Placebo — Sterile isotonic solution, subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a first-in-human, randomized, double-blind, placebo-controlled clinical study to evaluate the Safety and Tolerability of SPOT-mRNA01 injection in healthy adult volunteers.

DETAILED DESCRIPTION:
SPOT-mRNA01 (collagen 1 alpha 1 (COL1A1) mRNA-loaded by Extracellular vesicles （EVs）) can induce collagen protein grafts in dermal tissue, thereby supplementing collagen and reducing wrinkle formation in collagen-depleted skin. Therefore, SPOTmRNA01 can provide a source of human collagen intradermally for cosmetic anti-aging use.

This is a first-in-human randomized, double-blind, placebo-controlled, single-dose, dose ascending, exploratory clinical study to evaluate the Safety and Tolerability of SPOT-mRNA01 administered by subcutaneous injection to healthy adult volunteers.

Biopsies will be used to detect the expression of collagen in the skin of the injection area.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 to 75 years inclusive at the time of informed consent.

Exclusion Criteria:

1. Any transient or chronic skin condition, disorder, or infection within 20 cm of the target areas before treatment that, in the opinion of the investigator, may confound study results.
2. History of laser treatment or chemical peels or any cosmetic anti-aging treatments to the target areas within six months of the study treatment.
3. History of surgical procedures to target areas, including removal of benign or malignant skin cancers that, in the opinion of the investigator, may confound study results.
4. Participant with a history of heavy smoking, alcohol or drug abuse or steroid treatment.
5. Pregnant or breast-feeding females.
6. History of anaphylaxis or allergic reactions to any constituent of the study product and/or local anesthetics, and/or history of severe abnormal drug reaction.
7. Those who have participated in clinical trials of other investigational drugs within 3 months before the study treatment.
8. Those who are not suitable for subcutaneous injection and biopsy.
9. Any condition that the investigator or primary physician believes may not be appropriate for participating the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-12 (Estimated); Primary Completion 2027-11-12 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of the frequency and severity of AEs caused by SPOT-mRNA01 | 3 months
  The investigator will collect a description of the events, time of onset and resolution, assessment of severity and causal relationship to SPOT-mRNA01.

SECONDARY OUTCOMES:
level of COL1A1 protein expression in local dermal tissue after subcutaneous injection of SPOT-mRNA01 | Days 4, 7 and 31
  Local collagen expression in injection area biopsy by ELISA detection
Assessment of skin thickness after subcutaneous injection of SPOT-mRNA01 | Days 4, 7 and 31
  Detecting local skin thickness in injection site biopsy by Masson trichrome stain.
Assessment of skin thickness after subcutaneous injection of SPOT-mRNA01 | Baseline and days 7， 15， 31， 61 and 91
  Detecting local skin thickness by Skin ultrasound.